CLINICAL TRIAL: NCT01751828
Title: Late-life Depression and Cerebral Perfusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was an initial unfunded pilot project stopped after similar studies were funded.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Warren Taylor, Associate Professor of Clinical Psychiatry, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 121648
Record Dates: First submitted 2012-12-12; First posted 2012-12-18 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline (Experimental): Open-label sertraline, 8 week trial, dosing from 50mg to 200mg daily.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline
  Other Names: Zoloft

SUMMARY:
The long-term goal is to determine if decreased blood flow to the brain (cerebral hypoperfusion) is predictive of antidepressant outcomes in late-life depression (LLD). Studies in younger adult report that successful antidepressant treatment is associated with increases in cerebral blood flow, with no change in blood flow being observed in nonresponders. Thus cerebral hypoperfusion may be a biomarker of poor response to antidepressants. In LLD, this may occur secondarily to underlying vascular disease. If LLD is characterized by cerebral hypoperfusion and it does have predictive power to identify individuals who will poorly respond to conventional antidepressants, this would support the study of interventions that improve cerebral perfusion and may improve antidepressant outcomes.

As an initial step in this research, this pilot study will utilize MRI to examine if resting blood flow deficits predict and persist with antidepressant nonremission in an elderly population. The rationale for this proposal is that it will guide the design and power requirements of a larger, definitive trial examining the relationship between cerebral perfusion and depression outcomes. Importantly, support for this mechanism being linked to LLD would also support studies examining the antidepressant efficacy of drugs that may improve cerebral perfusion.

The primary purpose of this pilot study is a) to demonstrate feasibility by recruiting, scanning, and treating depressed elders; and b) to acquire preliminary data for competitive grant submissions.

SPECIFIC AIM: To use MRI to test for differences in cerebral perfusion between individuals who do and do not remit to a 8-week course of sertraline.

DETAILED DESCRIPTION:
After providing informed consent, participants will complete brain MRI and memory testing. If they are currently taking an antidepressant and are not doing well on it, they will be taken off it. Participants will then start sertraline, a commercially available antidepressants. They will be monitored for response and side effects for 8 weeks and doses adjusted as needed. After the study, we will examine how differences in brain blood flow may predict who does and does not respond to sertraline.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older.
* Current diagnosis of major depressive disorder (DSM-IV-TR), recurrent or chronic, without psychotic features
* Minimum depression severity of Montgomery Asberg Depression Rating Scale (MADRS) score ≥ 15
* Cognitively intact by Montreal Cognitive Assessment (MoCA) score ≥ 23
* Ability to read and write English

Exclusion Criteria:

* Other current or past psychiatric diagnoses
* Any use of illicit substances or abuse of prescription medications
* Presence of acute suicidality
* Current or past psychotic symptoms
* Known primary neurological disorder, including dementia
* Chronic untreated medical disorders where treatment is warranted
* Any contraindication to MRI, such as metal in the body
* Electroconvulsive therapy in the last 6 months
* Use of antidepressants or other psychiatric medications in the last month.
* Known allergy to sertraline
* A failed therapeutic trial of sertraline in the current depressive episode
* Current or planned psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 8 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms (QIDS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD, MHSc, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States